CLINICAL TRIAL: NCT02986711
Title: Pilot Randomized Trial of Brief Automated Smoking Cessation Intervention and Evaluation for Smokers Discharged From Hospital
Brief Title: Penn State TXT2STAYQUIT Study- a Texting Study to Help Hospitalized Smokers Stay Quit
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding exhausted
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Foulds, Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 40683
Record Dates: First submitted 2015-10-08; First posted 2016-12-08 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Nicotine Dependence, Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Text Messages (Experimental): Motivational text messages to help participants stay quit when they leave the hospital.
  Interventions: Behavioral: Motivational Text Messages
- Control (Sham Comparator): Text messages to ask about current smoking status.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Motivational Text Messages — Motivational text messages in addition to survey questions about smoking status
  Arms: Motivational Text Messages
Behavioral: Control — Only survey questions about smoking status
  Arms: Control

SUMMARY:
This study aims to pilot a method of collecting the post-discharge follow-up data required by the Joint Commission Tobacco Measure Set, using text messages sent to and received from patients' cellular-telephones. It also aims to assess whether specially designed relapse prevention text messages designed to encourage abstinence from smoking, can increase the proportion of smokers who remain abstinent during the first month after discharge from hospital.

DETAILED DESCRIPTION:
Participants will be those who are hospitalized at Hershey Medical Center and are interested in help to stay quit when they leave the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Total length of hospital stay at least 24 hours
* Free of cognitive impairment
* Read and speak English
* Smoked at least 20 cigarettes in 30 days prior to entering the hospital
* Willing to give up all forms of tobacco
* Has a cell phone capable of receiving text messages (cell phone is powered on and charged)

Exclusion Criteria:

* Patient has been admitted for a transplant
* Patient has Intensive Care status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Foulds, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivational Text Messages | Control
Started | 78 | 80
Completed | 70 | 70
Not Completed | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Text Messages | Control | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (13.3) | 42.5 (13.3) | 41.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 40 | 84
  Male | 26 | 30 | 56

OUTCOME MEASURES:

1. Primary Outcome: Complete Self-reported Tobacco Abstinence During the Prior 7 Days, as Reported on Telephone Interview, 28 Days After Discharge From Hospital (With Biochemical Verification in a Sub-sample, Exhaled Carbon-monoxide < 10 Parts Per Million).
Description: Abstinence rate at 28 days
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Text Messages | Control
Number analyzed (Participants) | 70 | 70
Participants | 31 | 26

2. Secondary Outcome: Proportion of Participants Providing Smoking Cessation Status Via Text Message
Description: proportion of participants providing data about smoking status via text message at 28 days
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Text Messages | Control
Number analyzed (Participants) | 70 | 70
Participants | 13 | 36

ADVERSE EVENTS:
Arm/Group | Motivational Text Messages | Control
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No